CLINICAL TRIAL: NCT00575237
Title: A Simple Clinical Maneuver to Reduce Laparoscopy Induced Shoulder Pain: A Randomized Clinical Trial
Brief Title: A Simple Clinical Maneuver to Reduce Laparoscopy Induced Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phelps, Paul, M.D. (Individual)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Phelps, Paul, M.D., Department of Anesthesia, Southwest Healthcare System, Murrieta, California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SP230819
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Shoulder Pain
Keywords: Laparoscopic Surgery; Shoulder pain; PDNV; Anesthesia; Residual CO2; Postoperative Pain; Female ASA 1 and 2 outpatients who were scheduled for elective gynecologic laparoscopic surgery
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): In the control group, CO2 was removed by passive deflation of the abdominal cavity through the holes of the trocar.
- Intervention (Experimental)
  Interventions: Procedure: Recruitment manouver

INTERVENTIONS:
Procedure: Recruitment manouver — In the intervention group, CO2 was removed by means of Trendelenburg position (> 30 degrees) with 5 manual pulmonary recruitment maneuvers.
  Arms: Intervention

SUMMARY:
A pulmonary recruitment maneuver at the end of surgery reduced shoulder pain as well as nausea and vomiting after laparoscopic surgery.

DETAILED DESCRIPTION:
With IRB approval and informed consent, 100 female ASA 1 and 2 outpatients who were scheduled for elective gynecologic laparoscopic surgery were randomly allocated to either the current standard (control group) or to additional efforts to remove residual CO2 at the end of surgery (intervention group; power analysis yielded 45 patients necessary per group). In the control group, CO2 was removed by passive deflation of the abdominal cavity through the holes of the trocar. In the intervention group, CO2 was removed by means of Trendelenburg position (> 30 degrees) with 5 manual pulmonary recruitment maneuvers. Postoperative shoulder pain was assessed prior to discharge and 12, 24, 36 and 48 hours later using a visual analog scale (VAS). In addition, positional characteristics of the shoulder pain and incidence of postdischarge nausea and vomiting (PDNV) were recorded 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 15-65
* ASA I-II
* scheduled for outpatient gynaecological procedure

Exclusion Criteria:

* previous laparatomy
* patients requiring hospitalisation
* procedure required conversion to laparatomy
* 48h follow-up no feasible

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-02; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Intensity of shoulder pain | 48 hours after discharge

SECONDARY OUTCOMES:
Incidence of Nausea and Vomiting | 24hrs after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Paul Phelps, MD, Principal Investigator — Department of Anesthesia, Southwest Healthcare System, Murrieta, California
Locations (1):
- Inland Valley and Rancho Springs Medical Centers, Wildomar, California, United States

REFERENCES:
- [Derived] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749